CLINICAL TRIAL: NCT03615716
Title: A Multi-level Approach to Violence Prevention Among African American
Brief Title: A Multi-level Approach to Violence Prevention Among African American Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Yu-Mei Schoenberger, Assistant Professor, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-300000551
Record Dates: First submitted 2018-07-09; First posted 2018-08-06 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Violence in Adolescence
Keywords: violence; adolescence

STUDY DESIGN:
Intervention Model Description: The study has 2 groups of participants. Only one group, middle school boys (N=20), will receive the intervention. But, pre- and post-assessments will be conducted with 2 groups: (1) boys, (2) caregivers. Caregivers (N=20) will give their perspectives of boys' behavior pre- and post- intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-level Violence Prevention Intervention - Boys (Experimental): A study examining middle school boys who have a high potential of violence based on where they live. This arm will measure outcomes in the boys. as the result of the intervention, from the perspectives of the boys.
  Interventions: Behavioral: Multi-level Violence Prevention Intervention - Boys
- Multi-level Violence Prevention Intervention - Caregivers (Experimental): In this study examining middle school boys who have a high potential of violence based on where they live, this arm will measure caregivers' perspectives of the boys ' outcomes. Caregivers will be surveyed pre-intervention and 4- and 6-month post intervention to explore the impact of the boys' intervention.
  Interventions: Behavioral: Multi-level Violence Prevention Intervention - Caregivers

INTERVENTIONS:
Behavioral: Multi-level Violence Prevention Intervention - Boys — Comprehensive, Multi-level Violence Prevention Intervention. The intervention consists of three components: (1) a 15-week after-school program, (2) group mentoring, and (3) community enhancement activities. Adolescents and mentors will attend a 2-hour weekly session at a community center, and will conduct up to four community enhancement activities. At the end of the program, a graduation celebration will be planned, and parents/guardians and stakeholders (e.g., coalition members) will be invited.
  Arms: Multi-level Violence Prevention Intervention - Boys
Behavioral: Multi-level Violence Prevention Intervention - Caregivers — This is arm is measuring the Multi-level Violence Prevention Intervention that is administered to the boys, from the perspectives of their caregivers. The caregivers themselves will not receive an intervention, but their perspectives of the impact on the interventions on the boys will be examined
  Arms: Multi-level Violence Prevention Intervention - Caregivers

SUMMARY:
The overall goal of this study is to advance the science of youth violence prevention and the social determinants of health by using a community-driven approach to implement a comprehensive intervention. The objective of the proposed project is to assess the feasibility, acceptability, and preliminary efficacy of an innovative, multi-level intervention that promotes adolescent protective factors and reduces risk behaviors among African American youth residing in Birmingham. Alabama.

DETAILED DESCRIPTION:
Perceived neighborhood violence, hearing about violence in one's community, and being a victim of violence contributes to adverse psychological conditions such as anxiety, depression, and stress, which may have cascading negative effects physically and be the start of a vicious cycle. Among children, the prevalence of neighborhood violent crime is linked to symptoms of post-traumatic stress disorder (PTSD), aggressive behavior, school attendance problems, sexual risk taking, and the use of alcohol, tobacco, and other drugs.

Since childhood is a critical and fragile time with respect to developmental trajectories and relationship building, it is an important time to intervene. Previous research used a deficit model focusing on risks as opposed to an asset model, which focuses on protective factors related to prosocial and positive traits. Building the protective factors (e.g., involvement in prosocial activities, intolerant attitude toward deviance, connectedness to adults outside the family) of youth can promote well-being and reduce the risks of negative outcomes. Social-emotional learning (SEL) programming targeting adolescents is thus becoming increasingly funded because of its documented success, such as higher levels of prosocial behavior, more favorable attitudes toward school and others, and better academic achievement.

The overall goal of this study is to advance the science of youth violence prevention and the social determinants of health by using a community-driven approach to implement a comprehensive intervention. The objective of the proposed project is to assess the feasibility, acceptability, and preliminary efficacy of an innovative, multi-level intervention that promotes adolescent protective factors and reduces risk behaviors among African American youth residing in Birmingham. Alabama. According to data from the FBI's 2015 Uniform Crime Report, Birmingham is ranked as the nation's 3rd most violent city with high levels of violent crime occurring in the a neighborhood located in Northeast Birmingham, Alabama. By partnering with national and local community partners, this study proposes to design a comprehensive intervention that integrates an evidence-based, individual-level SEL program with a relationship-level mentoring component and a community-level environmental improvement component. The proposed pilot project is building on recently established community relationships. Through community capacity development funds, the investigators helped establish a community coalition in Spring of 2016 to identify and address the underlying causes of health disparities in the community. The coalition has identified violence and safety as issues that community members most desire to be addressed and has recommended strategies, such as establishing a mentoring program, providing activities for children, and organizing community improvement activities. The proposed project addresses several of these issues and our community partners have expressed enthusiastic support of the project.

The proposed project will be achieved through the following specific aims:

Aim 1: Conduct a 4-month multi-level youth violence prevention intervention that includes an individual-level social-emotional learning program with a relationship-level mentoring component and a community-level environmental improvement component. The intervention will include 20 African American male adolescents residing in a community in Birmingham, AL.

Aim 2: Assess the feasibility and acceptability of the multi-level intervention.

1. Feasibility and Acceptability (Primary Outcome): Detailed process data will be collected to assess recruitment, retention, and acceptance. It is hypothesized that 20 African American adolescents (6th-8th grade) will be recruited, >80% of the participants will be retained, and >80%will accept the intervention.
2. Efficacy (Secondary Outcome): To determine the effects of the intervention on aggressive behavior and prosocial behavior (protective factors). It is hypothesized that participants will have significantly lower levels of aggressive behavior and higher levels of prosocial behavior.

This study will be a significant contribution to the multi-level violence prevention literature and lay the foundation for a larger study using an experimental design to examine effects of a violence prevention intervention on individual and community health and well-being. In addition, lessons learned from this project can serve as a model to address violence prevention in similar inner-city communities in the United States.

ELIGIBILITY:
Boys Inclusion Criteria:

* Male
* Identify as African American or Black
* aged 11-14 years at the time of the study enrollment
* Reside in the targeted community
* Be able to meet after school once a week for 4-months.

Boys Exclusion Criteria:

* Not English speaking

Caregivers Inclusion Criteria:

* Identify as the primary caregiver of a boy enrolled in the study

Caregivers Exclusion Criteria:

* Not English speaking

Ages: 11 Years to 14 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 32 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2019-06-12 (Actual)

PRIMARY OUTCOMES:
Evaluate behavior using the Strengths and Difficulties Questionnaire | At baseline
  25-item self-report Strengths and Difficulties Questionnaire (SDQ) validated for ages 11-16. It is divided into 5 scales: emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behavior (α=.73)
Evaluate behavior using the Strengths and Difficulties Questionnaire | From baseline through 4 months
  25-item self-report Strengths and Difficulties Questionnaire (SDQ) validated for ages 11-16. It is divided into 5 scales: emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behavior (α=.73)
Evaluate behavior using the Strengths and Difficulties Questionnaire | From baseline through 6 months
  25-item self-report Strengths and Difficulties Questionnaire (SDQ) validated for ages 11-16. It is divided into 5 scales: emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behavior (α=.73)
Child aggressive behavior and prosocial skills - for parent/guardian to complete | baseline
  25-item parent Strengths and Difficulties Questionnaire (SDQ) measures child's behavior from parent perspective. It is divided into 5 scales: emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behavior.
Child aggressive behavior and prosocial skills - for parent/guardian to complete | 4 months
  25-item parent Strengths and Difficulties Questionnaire (SDQ) measures child's behavior from parent perspective. It is divided into 5 scales: emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behavior.
Child aggressive behavior and prosocial skills - for parent/guardian to complete | 6 months
  25-item parent Strengths and Difficulties Questionnaire (SDQ) measures child's behavior from parent perspective. It is divided into 5 scales: emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behavior.

SECONDARY OUTCOMES:
Perceived Satisfaction | 4 months
  6-item intervention satisfaction measure
Participant satisfaction with mentors | 4 months
  adaptation of a satisfaction with patient navigator questionnaire
Utilization - Sessions | 4 months
  number of sessions attended
Utilization - community service activities | 4 months
  number of community activities attended
Utilization - time with mentor | 4 months
  total minutes spent with mentor
Sense of Belonging Scale | baseline
  5-item 5-point likert scale measures sense of belonging in the program (i.e., connected, committed, supported, accepted). Validated among ages 9-19 (α=.93).
Sense of Belonging Scale | 4 months
  5-item 5-point likert scale measures sense of belonging in the program (i.e., connected, committed, supported, accepted). Validated among ages 9-19 (α=.93).
Sense of Belonging Scale | 6 months
  5-item 5-point likert scale measures sense of belonging in the program (i.e., connected, committed, supported, accepted). Validated among ages 9-19 (α=.93).
School Safety | baseline
  1-item 5-point likert scale assessing agreement with the statement, "I feel safe at my school" (strongly agree to strongly disagree). Has been shown to have validity and reliability in terms of both predictors (e.g., sociodemographics) and predicting outcomes (e.g., well-being).
School Safety | 4 months
  1-item 5-point likert scale assessing agreement with the statement, "I feel safe at my school" (strongly agree to strongly disagree). Has been shown to have validity and reliability in terms of both predictors (e.g., sociodemographics) and predicting outcomes (e.g., well-being).
School Safety | 6 months
  1-item 5-point likert scale assessing agreement with the statement, "I feel safe at my school" (strongly agree to strongly disagree). Has been shown to have validity and reliability in terms of both predictors (e.g., sociodemographics) and predicting outcomes (e.g., well-being).
Neighborhood safety | baseline
  4-item 5-point likert scale includes items such as "It's safe to walk around my neighborhood" and "I'm scared of people in my neighborhood" with higher scores indicating greater neighborhood safety (α=.77).
Neighborhood safety | 4 months
  4-item 5-point likert scale includes items such as "It's safe to walk around my neighborhood" and "I'm scared of people in my neighborhood" with higher scores indicating greater neighborhood safety (α=.77).
Neighborhood safety | 6 months
  4-item 5-point likert scale includes items such as "It's safe to walk around my neighborhood" and "I'm scared of people in my neighborhood" with higher scores indicating greater neighborhood safety (α=.77).
Neighborhood Cohesion | baseline
  5-item 5-point likert scale measuring how much they agree with statements regarding their neighborhood and neighbors such as "people in this neighborhood can be trusted," "people in this neighborhood do not share the same values," and "there are people I can count on in this neighborhood."
Neighborhood Cohesion | 4 months
  5-item 5-point likert scale measuring how much they agree with statements regarding their neighborhood and neighbors such as "people in this neighborhood can be trusted," "people in this neighborhood do not share the same values," and "there are people I can count on in this neighborhood."
Neighborhood Cohesion | 6 months
  5-item 5-point likert scale measuring how much they agree with statements regarding their neighborhood and neighbors such as "people in this neighborhood can be trusted," "people in this neighborhood do not share the same values," and "there are people I can count on in this neighborhood."
Family Cohesion | baseline
  12-item subscale contains items related to family communication and closeness.
Family Cohesion | 4 months
  12-item subscale contains items related to family communication and closeness.
Family Cohesion | 6 months
  12-item subscale contains items related to family communication and closeness.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Mei Schoenberger, PhD, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- The University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/16/NCT03615716/ICF_000.pdf